CLINICAL TRIAL: NCT00125684
Title: Bioavailability and Effectiveness of Transdermally Administered Morphine
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Alberta Health services (Other)
Collaborators: Tom Baker Cancer Centre (Other)
Responsible Party: Principal Investigator, Rachel Syme, Dr. Neil Hagen - Principal Investigator, Alberta Health services
Organization: AHS Cancer Control Alberta (Other)
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 10181
Record Dates: First submitted 2005-07-29; First posted 2005-08-02 (Estimated); Last update posted 2012-01-19 (Estimated); Status verified 2011-08

CONDITIONS: Cancer; Pain
Keywords: transdermal morphine; cancer; pain; bioavailability; pharmacokinetics; cancer related pain; stable baseline pain; currently taking opioids
MeSH Terms: conditions — Neoplasms; Pain; Cancer Pain | interventions — Morphine

INTERVENTIONS:
Drug: morphine

SUMMARY:
Patients will participate in two arms of the trial, one in which morphine will be administered transdermally, and, after a 3 day wash out period, one in which morphine will be administered subcutaneously.

DETAILED DESCRIPTION:
Patients will participate in two arms of the trial, one in which morphine will be administered transdermally, and, after a 3 day wash out period, one in which morphine will be administered subcutaneously. Blood draws will be done after both dosing methods in order to compare blood levels of morphine by the different routes.

ELIGIBILITY:
Inclusion Criteria:

* Chronic cancer pain
* Minimum baseline pain of 3/10
* No change in medications over 3 days prior to study period
* Ability to give informed consent
* Willingness to undergo repeated blood sampling

Exclusion Criteria:

* Use of morphine or codeine in 3 days prior to study
* Known sensitivity to morphine
* Prior anaphylactic reaction to any opioid
* Clinically significant anemia

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 6 (Estimated)
Dates: Start 2003-07; Primary Completion 2007-07 (Actual); Study Completion 2008-07 (Actual)

PRIMARY OUTCOMES:
detectable morphine levels in serum

CONTACTS AND LOCATIONS:
Overall Officials: Neil Hagen, Principal Investigator — Alberta Cancerboard
Locations (1):
- Tom Baker Cancer Centre, Calgary, Alberta, Canada